CLINICAL TRIAL: NCT02526537
Title: The Postoperative Adjuvant Therapy of Gefitinib for High Risk Stage Ib NSCLC Patients With EGFR Sensitive Mutation, an Open, Paired, Non-interventional, Multi-center Clinical Study
Brief Title: Gefitinib for EGFR Sensitive Mutation Postoperative Stage Ib NSCLC Patients
Status: Terminated | Type: Observational
Why Stopped: Similar study has revealed result of no benefit for participants
Sponsor: Lunxu Liu (Other)
Responsible Party: Sponsor-Investigator, Lunxu Liu, chief physician, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: TSCI001
Record Dates: First submitted 2015-08-11; First posted 2015-08-18 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: NSCLC
Keywords: Gefitinib; NSCLC; postoperative; stage Ib; Relapse Free Survival in 2 years

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Gefitinib: Stage IB NSCLC Patients with high risk factors and EGFR gene sensitive mutation who can not tolerate or decline chemotherapy and choose Gefitinib for postoperative therapy (Gefitinib 250 mg daily for 2 years).
- Non-specific treatment: Stage IB NSCLC Patients with high risk factors and EGFR gene sensitive mutation who can not tolerate or decline chemotherapy and choose Non-specific treatment.(Chinese herbal medicine and nonspecific immunomodulators as adjuvant anti-cancer treatment for 2 years).

SUMMARY:
Currently, whether adjuvant therapy should be applied to Stage Ib non-small cell lung cancer (NSCLC) patients who received radical resection remains controversial. There is still no clear evidence that the postoperative adjuvant chemotherapy or other treatments can improve the survival rate for patients with stage Ib NSCLC. Tyrosine Kinase Inhibitors (TKIs) such as Gefitinib and Erlotinib are widely accepted as the first-line therapy for Epidermal growth factor receptor (EGFR) gene mutation late stage NSCLC patients. However the effect is largely uncertain for early stage patients who received surgery. The investigators aim to evaluate the effect of postoperative adjuvant use of Gefitinib for high risk stage Ib EGFR sensitive mutation NSCLC patients.

DETAILED DESCRIPTION:
Currently, whether adjuvant therapy should be applied to Stage Ib non-small cell lung cancer (NSCLC) patients who received radical resection remains controversial. CALGB9633 studies have shown that for patients with stage Ib NSCLC who received radical resection, postoperative adjuvant chemotherapy does not benefit for all patients, only patients with high risk (cancer diameter >4cm) can benefit. There is still no clear evidence that the postoperative adjuvant chemotherapy or other treatments can improve the survival rate for patients with stage Ib NSCLC.

The EGFR gene mutation rate is about 10% for European patients, and about 30-40% for patients of Asian origins. In a retrospective observation study of 1118 stage I to stage III NSCLC patients who received surgery, D'Angelo et al. found that the risk of death for patients with EGFR sensitive mutation is lower than those without mutation. The authors indicated that postoperative use of TKI for EGFR sensitive mutation patients might be the possible reason. Since the mutation rate of EGRF gene is higher in Asian patients, compared with patients of other origins, the investigators speculate that Asian patients might benefit for postoperative use of TKIs.

EGFR gene mutation detection is routinely prescribed nowadays for lung adenocarcinoma patients who received surgical resection. According to NCCN guideline, stage IB patients with high risk factors are recommended to receive adjuvant chemotherapy. For patients who can not tolerate or decline chemotherapy, non-specific treatment ( Chinese herbal medicine and nonspecific immunomodulators as adjuvant anti-cancer treatment for 2 years) is recommended, otherwise, TKIs（Gefitinib 250 mg daily for 2 years) is also an alternative choice if the cancer has EGFR sensitive mutation. Based on patient's own choice of postoperative adjuvant therapy , the patients were enrolled for observation of prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. High-risk who meet one of the following descriptions: 1). Poorly differentiated carcinoma (including neuroendocrine tumors); 2). Vascular invasion; 3). Tumor diameter≥4cm 5). Visceral pleura involvement.
2. Patients with pathology confirmed Ib stage NSCLC
3. Patients with deletion of exon 19 or mutation of L858R at exon 21 in EGFR gene
4. ECOG score of 0-1
5. Life expectancy over 12 weeks
6. Absolute neutrophil count (ANC) >= 1.75 x 109 / L, platelet >= 100 x 109 / L, hemoglobin is more than or equal to 9 g / dl
7. Total bilirubin <= the normal value of 1.5 times the upper limit of normal (ULN); liver metastases, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) <= 2.5 times of upper limit of normal (ULN)
8. Serum creatinine <=1.25 times of the upper limit of normal value, creatinine clearance rate > 60 or ml/min
9. received the informed consent from patient or his/her legal representative

Exclusion Criteria:

1. Patients who was serious allergy to any of the ingredients of drugs used in this study
2. Patients who unable to comply with the study plan or research program;
3. Patients with severe systemic disease that the researchers judged will be unable to complete the study;
4. Patients have severe heart disease, such as myocardial infarction within 6 months;
5. Patients have interstitial pneumonia;
6. Patients who were confirmed to be positive pathology for cutting edge;
7. The preoperative chest CT showed nodules >= 50%, and showed ground glass opacity;
8. Patients received wedge resection;
9. Patients used HER2 pathways involved drugs such as erlotinib, gefitinib, cetuximab rituximab, trastuzumab)
10. Patients who have received chemotherapy or systemic antitumor therapy (such as monoclonal antibody therapy);
11. Patients received radiotherapy;
12. Having other malignant tumors in the last 5 years, but not including who has been cured through surgery and survived 5 year of disease-free;
13. Any unstable systemic diseases (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, or myocardial infarction, serious arrhythmias, liver, kidney or metabolic diseases within six months).
14. Patients who do not get effective treatment of inflammation, eye infections or predisposing factors;
15. Physical examination or laboratory findings evidence reasonable doubt who is ill or use of related drugs could affect the study;
16. Patients with serious active infections;
17. Patients with T790M mutations at 20 exon;
18. Woman who are pregnant or lactating.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients received complete resection at stage Ib with deletion of exon 19 or mutation of L858R at exon 21 in EGFR
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-11-11 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Relapse Free Survival in 2 years | Treatment period: 2 years (24 months)

SECONDARY OUTCOMES:
Relapse Free Survival in 3 years | Follow-up: 3 years
5 year Overall Survival | Follow-up: 5 years
Relapse Free Survival in 5 years | Follow-up: 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lunxu Liu, Professor, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Wu YL, Zhong WZ, Li LY, Zhang XT, Zhang L, Zhou CC, Liu W, Jiang B, Mu XL, Lin JY, Zhou Q, Xu CR, Wang Z, Zhang GC, Mok T. Epidermal growth factor receptor mutations and their correlation with gefitinib therapy in patients with non-small cell lung cancer: a meta-analysis based on updated individual patient data from six medical centers in mainland China. J Thorac Oncol. 2007 May;2(5):430-9. doi: 10.1097/01.JTO.0000268677.87496.4c. PMID 17473659
- [Background] Strauss GM, Herndon JE 2nd, Maddaus MA, Johnstone DW, Johnson EA, Harpole DH, Gillenwater HH, Watson DM, Sugarbaker DJ, Schilsky RL, Vokes EE, Green MR. Adjuvant paclitaxel plus carboplatin compared with observation in stage IB non-small-cell lung cancer: CALGB 9633 with the Cancer and Leukemia Group B, Radiation Therapy Oncology Group, and North Central Cancer Treatment Group Study Groups. J Clin Oncol. 2008 Nov 1;26(31):5043-51. doi: 10.1200/JCO.2008.16.4855. Epub 2008 Sep 22. PMID 18809614
- [Background] D'Angelo SP, Janjigian YY, Ahye N, Riely GJ, Chaft JE, Sima CS, Shen R, Zheng J, Dycoco J, Kris MG, Zakowski MF, Ladanyi M, Rusch V, Azzoli CG. Distinct clinical course of EGFR-mutant resected lung cancers: results of testing of 1118 surgical specimens and effects of adjuvant gefitinib and erlotinib. J Thorac Oncol. 2012 Dec;7(12):1815-1822. doi: 10.1097/JTO.0b013e31826bb7b2. PMID 23154553
- [Background] Tsuboi M, Kato H, Nagai K, Tsuchiya R, Wada H, Tada H, Ichinose Y, Fukuoka M, Jiang H. Gefitinib in the adjuvant setting: safety results from a phase III study in patients with completely resected non-small cell lung cancer. Anticancer Drugs. 2005 Nov;16(10):1123-8. doi: 10.1097/00001813-200511000-00012. PMID 16222155
- [Background] Janjigian YY, Park BJ, Zakowski MF, Ladanyi M, Pao W, D'Angelo SP, Kris MG, Shen R, Zheng J, Azzoli CG. Impact on disease-free survival of adjuvant erlotinib or gefitinib in patients with resected lung adenocarcinomas that harbor EGFR mutations. J Thorac Oncol. 2011 Mar;6(3):569-75. doi: 10.1097/JTO.0b013e318202bffe. PMID 21150674
- [Background] Zhang Shunda, Deng Yanming, Feng Weineng, Chen Zecheng. Clinical Effects of Gefitinib Tablets in Auxiliary Treatment of Non-small Cell Lung Cancer and its Influencing Factors. Anti-tumor Pharmacy2013, 3(4): 278-281.
- [Background] Goss GD, O'Callaghan C, Lorimer I, Tsao MS, Masters GA, Jett J, Edelman MJ, Lilenbaum R, Choy H, Khuri F, Pisters K, Gandara D, Kernstine K, Butts C, Noble J, Hensing TA, Rowland K, Schiller J, Ding K, Shepherd FA. Gefitinib versus placebo in completely resected non-small-cell lung cancer: results of the NCIC CTG BR19 study. J Clin Oncol. 2013 Sep 20;31(27):3320-6. doi: 10.1200/JCO.2013.51.1816. Epub 2013 Aug 26. PMID 23980091
- [Background] Li N, Ou W, Ye X, Sun HB, Zhang L, Fang Q, Zhang SL, Wang BX, Wang SY. Pemetrexed-carboplatin adjuvant chemotherapy with or without gefitinib in resected stage IIIA-N2 non-small cell lung cancer harbouring EGFR mutations: a randomized, phase II study. Ann Surg Oncol. 2014 Jun;21(6):2091-6. doi: 10.1245/s10434-014-3586-9. Epub 2014 Mar 1. PMID 24585406